CLINICAL TRIAL: NCT06856434
Title: Effect of Consumption of Lactobacillus Plantarum Sp Probiotics on Leukocyte Levels, Segment Neutrophil Type Counts, Post-operative Pain, and Length of Stay in Patients with Diffuse Peritonitis Due to the Perforated Appendix That Has Been Performed Laparotomy Appendectomy At Dr. Hasan Sadikin Hospital: a Randomized Controlled Trials
Brief Title: Effect of Probiotic's Consumption on Several Markers in Perforated Appendix Patients with Diffuse Peritonitis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Ricarhdo Valentino Hanafi, MD, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SURG-202407.01
Record Dates: First submitted 2025-02-20; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Appendicitis with Perforation; Appendectomy; Probiotic
Keywords: Perforated Appendicitis; Appendectomy; Probiotic; Laparotomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic Group (Experimental): Patient with perforated appendicitis who received an intervention
  Interventions: Dietary Supplement: Lactobacillus plantarum sp Probiotic
- Placebo Group (Placebo Comparator): Patients with perforated appendicitis who did not receive an intervention
  Interventions: Other: Placebo Group

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum sp Probiotic — Once daily consumption
  Arms: Probiotic Group
Other: Placebo Group — Group who received a placebo intervention
  Arms: Placebo Group

SUMMARY:
Does the administration of the probiotic Lactobacillus plantarum sp. have an impact on reducing leukocyte levels, segmented neutrophil counts, postoperative pain, and length of hospitalization in patients with diffuse peritonitis caused by perforated acute appendicitis who underwent laparotomy appendectomy at Dr. Hasan Sadikin Hospital?

DETAILED DESCRIPTION:
To determine whether the administration of the probiotic Lactobacillus plantarum sp. to patients with diffuse peritonitis caused by appendiceal perforation undergoing laparotomy appendectomy at Hasan Sadikin Hospital Bandung and Siloam Karawaci Hospital has a significant effect on leukocyte levels, segmented neutrophil counts, postoperative pain levels, and length of hospitalization compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diffuse peritonitis caused by appendicitis
* Patients undergoing laparotomic appendectomy.
* Patients aged 18 years or older.

Exclusion Criteria:

* Patients with a history of previous laparotomy.
* Patients who underwent laparotomy combined with surgery on other parts of the body.
* Patients with a history of cancer.
* Patients with pre-existing comorbidities (uncontrolled diabetes mellitus, congestive heart failure, end-stage renal disease [ESRD], human immunodeficiency virus [HIV], and systemic lupus erythematosus [SLE]).
* Patients with multiple organ dysfunction syndrome (MODS).
* Patients with prior consumption of probiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
White Blood Cells Level | From the day of randomization up to 5 days postoperatively
  A white blood count measures the number of white blood cells (WBCs) in patients' blood.

SECONDARY OUTCOMES:
Segmented Neutrophil level | From the day of randomization up to 5 days postoperatively
  Segmented neutrophils are the most mature neutrophilic granulocytes present in circulating blood
Post operative pain level | From the day of randomization up to 5 days postoperatively
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'
Length of Hospital Stay | From the day of randomization up to 5 days postoperatively
  The duration of a single episode of hospitalization

IPD SHARING:
Plan to Share IPD: Yes
All data will be available for public
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Guan L, Liu Z, Pan G, Zhang B, Wu Y, Gan T, Ouyang G. The global, regional, and national burden of appendicitis in 204 countries and territories, 1990-2019: a systematic analysis from the Global Burden of Disease Study 2019. BMC Gastroenterol. 2023 Feb 22;23(1):44. doi: 10.1186/s12876-023-02678-7. PMID 36814190